CLINICAL TRIAL: NCT04780711
Title: Prevalance of Temporomandibular Joint Disease in Medical School Students
Brief Title: Prevalance of Temporomandibular Joint Disease
Status: Completed | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Elif yaksi, Medical Doctor, Abant Izzet Baysal University
Other Study IDs: AIBU-FTR-EY-01
Record Dates: First submitted 2021-02-21; First posted 2021-03-03 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Temporomandibular Joint Disorders
Keywords: Temporomandibular Joint Disorders
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diagnostic Group: Demographic data, symptoms for TMJ of the students will be recorded. Physical examination will be included range of motion of temporomandibular joint, right and left TMJ lateral range of motion, whether there is a gradual opening, during deflection and deviation during the opening and subluxation for palpation and measurements. Opening and closing clicks, crepitation and popping will be recorded during palpation. Deep palpation of the skin, masseter and temporal muscles will be determined, posture analysis will be recorded and dental interventions, missing teeth, orthodontic treatments and bruxism histories will be taken. An appropriate diagnosis will be determined for students who are found to have pathology as a result of all these examinations and information about this diagnosis will be provided.

SUMMARY:
Temporomandibular joint (TMJ) disorders are common problems in the society and involve the masticator muscles, jaw joint and related structures. Since TMJ disorders affect functions such as eating and speaking, they can cause important problems in the daily life of the patient. Therefore, its diagnosis and treatment are of great importance. In the treatment of these patients, methods such as analgesic and anti-inflammatory drugs, splint, exercise, physical therapy modalities can be applied.

DETAILED DESCRIPTION:
Although the prevalence of TMJ disease detected in the community is between 40-60%, the rate of symptoms or clinical findings was reported to be 87% in a study including 1040 people. Incomplete clarification of the etiology and pathogenesis, the lack of standard diagnostic and treatment approaches cause patients to learn to live with this problem, and severe pain and limitation of movement cause a decrease in quality of life and loss of workforce. Specific pathologies such as systemic inflammatory diseases, tumor, fracture, developmental anomaly cause temporomandibular joint diseases. It also causes a wider group of non-specific TMB originating from the musculoskeletal system.When the literature was reviewed, no publications on the frequency of TMJ joint disease were found in medical faculty students.

ELIGIBILITY:
Inclusion Criteria:

* Being a medical student
* Being between the ages of 18-35

Exclusion Criteria:

* Students who do not want to participate in the study

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: We planned to include 500 volunteer students between the ages of 18-35, studying at Bolu Abant Izzet Baysal University Faculty of Medicine, with or without TMJ symptoms and agreeing to participate in the study.
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2021-03-20 (Actual); Primary Completion 2021-07-28 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Mouth opening | Baseline
  The patient opens her mouth to the maximum, the lower border of the anterior upper teeth and the distance to the upper border of the lower teeth are measured.
Tenderness in the masseter and temporal muscles on deep palpation | Baseline
  Tenderness in the masseter and temporal muscles on deep palpation
Click in the temporomandibular joint | Baseline
  The patient's temporomandibular joint is palpated, and it is checked whether there is click or popping when opening or closing the mouth.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Yakşi, MD, Principal Investigator — Abant İzzet Baysal University Medical Faculty
Locations (1):
- Elif Yakşi, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No